CLINICAL TRIAL: NCT02638623
Title: Does Fluid Replacement From Preoperative NPO Status Improve Postoperative Recovery and Reduce Complications in Arthroplasty Patients?
Brief Title: Does Fluid Replacement From Preoperative NPO Status Improve Postoperative Recovery
Acronym: Hydration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Matthew Dietz, MD, Assistant Professor, MD, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1502590723
Record Dates: First submitted 2015-12-18; First posted 2015-12-23 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis
Keywords: Knee Arthroplasty; Hip Arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Ringer's Lactate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Lactated Ringer (Active Comparator): Covered two liters of body temperature warmed lactated ringer's in the immediate preoperative setting of subjects undergoing total knee or total hip replacement
  Interventions: Drug: Lactated Ringer
- Placebo (Placebo Comparator): Covered empty bag with no hydration supplement
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactated Ringer — 2L Lactated Ringer administered prior to primary knee or hip arthroplasty
  Arms: Drug Lactated Ringer
Drug: Placebo — No additional fluids will be administered
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The investigators are testing the hypothesis that administering 2L of body temperature warmed lactated ringer's intravenously prior to surgery can optimize the postoperative and recovery of patients undergoing total hip and total knee arthroplasty.

DETAILED DESCRIPTION:
Hip and knee arthroplasty are safe and reliable surgeries for the majority of patients, but a small percentage experience major complications such as myocardial infarction, deep vein thrombosis (DVT), and pulmonary embolism (PE). As these complications are related to local tissue hypoxemia and patient immobility, interventions that can improve the ability of the heart to deliver blood to the tissue and help patients mobilize earlier in their postoperative course may decrease these complications. Based on recent evidence, it has been shown that many patients are dehydrated before surgery, which can make them feel nauseous, tired, and increase their perception of pain making them less likely to mobilize. This predisposes them to DVTs, pulmonary embolism, nausea and vomiting. Peri-operative dehydration can also decrease the ability of the lungs to oxygenate the blood properly and can place additional stress on the heart, which can increase the risk of heart attacks. The specific aim is to determine if patients' peri-operative hemodynamics can be improved with preoperative administration of 2 L of lactated ringers, and consequently reduce postoperative complications and improve recovery in arthroplasty patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients >= 18 years of age, undergoing a total primary knee or hip arthroplasty

Exclusion Criteria:

* Patients weighing less than 80 kg.
* Patients undergoing irrigation and debridement, explantation, or revision will not be eligible.
* history of kidney disease, congestive heart failure, pulmonary edema, cirrhosis of the liver, or history of systemic fluid overloard will be excluded from the study.
* No one will be excluded based on gender, ethnicity or race.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Dietz, MD, Principal Investigator — West Virginia University Department of Orthopaedics
Locations (1):
- WVU Medicine Department of Orthopaedics, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lactated Ringer Bolus Group: Covered two liters of body temperature warmed lactated ringer's in the immediate preoperative setting of subjects undergoing total knee or total hip replacement
  Lactated Ringer: 2L Lactated Ringer administered prior to primary knee or hip arthroplasty
Period: Overall Study
Arm/Group | Lactated Ringer Bolus Group | Placebo
Started | 27 | 25
Completed | 20 | 19
Not Completed | 7 | 6
Not completed — Surgery timing | 5 | 6
Not completed — Not given intervention | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactated Ringer Bolus Group | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants] — Population: 52 participants were initially enrolled. Patients that did not have surgery were removed from the analysis. Also, there were a few instances where there was not adequate staffing to fulfill the protocols needs.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 19 | 14 | 33
    >=65 years | 1 | 5 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 52 participants were initially enrolled. Patients that did not have surgery were removed from the analysis. Also, there were a few instances where there was not adequate staffing to fulfill the protocols needs.
  Participants
    Female | 12 | 5 | 17
    Male | 8 | 14 | 22
Region of Enrollment [Number; unit: participants] — Population: 52 participants were initially enrolled. Patients that did not have surgery were removed from the analysis. Also, there were a few instances where there was not adequate staffing to fulfill the protocols needs.
  participants
    United States | 20 | 19 | 39
Surgical Procedure [Count of Participants; unit: Participants] — Population: 52 participants were initially enrolled. Patients that did not have surgery were removed from the analysis. Also, there were a few instances where there was not adequate staffing to fulfill the protocols needs.
  Participants
    Hip Replacement | 4 | 11 | 15
    Knee Replacement | 16 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Complications
Description: Patients found to have a 90-day postoperative complication categorized as Infection, CHF/Fluid overload, MI, DVT/PE, other
Time Frame: 90 days post surgery
Population: Chart review for patients up to 90 days after surgery documenting the above complications.
Measure: Number; unit: participants
Arm/Group | Lactated Ringer Bolus Group | Placebo
Number analyzed (Participants) | 20 | 19
participants
  Wound Infection | 0 | 1
  DVT/PE | 0 | 0
  MI | 0 | 0
  CHF/Fluid Overload | 0 | 0
  Other | 2 | 0

2. Secondary Outcome: 90 Day Readmission Count
Description: Patient readmitted to the hospital 90 day postoperatively
Time Frame: 90 days postop
Measure: Count of Participants; unit: Participants
Arm/Group | Lactated Ringer Bolus Group | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Readmission | 0 | 1
  No Readmission | 20 | 18

3. Secondary Outcome: Duration of Hospital Stay (Hours)
Description: Hours of Hospital Stay
Time Frame: Surgery to hospital discharge
Measure: Mean (Full Range); unit: hours
Arm/Group | Lactated Ringer Bolus Group | Placebo
Number analyzed (Participants) | 20 | 19
hours | 53.86 [26 to 169] | 36.13 [24 to 78]

4. Secondary Outcome: Duration of Surgery
Description: Minutes recorded for length of surgery
Time Frame: Incision to end of surgery
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Lactated Ringer Bolus Group | Placebo
Number analyzed (Participants) | 20 | 19
Minutes | 122.68 [87 to 172] | 126.3 [102 to 158]

5. Secondary Outcome: Emesis Episodes
Description: Number of recorded emesis episodes in the medical record while patient was hospitalized
Time Frame: Hospital Stay
Measure: Mean (Full Range); unit: emesis episodes
Arm/Group | Lactated Ringer Bolus Group | Placebo
Number analyzed (Participants) | 20 | 19
emesis episodes | 0.26 [0 to 2] | 0.11 [0 to 1]

6. Secondary Outcome: Volume of Fluid Administred
Description: milliliters of fluid administered during surgery
Time Frame: surgical period
Measure: Mean (Full Range); unit: milliliters
Arm/Group | Lactated Ringer Bolus Group | Placebo
Number analyzed (Participants) | 20 | 19
milliliters | 1635 [400 to 4750] | 1518 [700 to 2600]

ADVERSE EVENTS:
Time Frame: 90 Days postoperatively
Arm/Group | Lactated Ringer Bolus Group | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No